CLINICAL TRIAL: NCT04462198
Title: A Phase I/IIa, Randomized, Double-Blind, Placebo-Controlled, Safety, Pharmacokinetic, and Preliminary Efficacy Study of Unilateral Intratympanic PIPE-505 in Subjects With Sensorineural Hearing Loss Associated With Speech-in-Noise Impairment
Brief Title: Phase I/IIa Study Evaluating Safety and Efficacy of an Intratympanic Dose of PIPE-505 in Subjects With Hearing Loss
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Contineum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTI-505-101
Record Dates: First submitted 2020-06-29; First posted 2020-07-08 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2020-10

CONDITIONS: Sensorineural Hearing Loss
Keywords: Hearing Loss; Cochlear synaptopathy; Deafness; Speech-in-noise hearing difficulty
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss; Hearing Loss, Hidden; Deafness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The dose preparer and treatment administrator will be unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PIPE-505 (Experimental)
  Interventions: Drug: PIPE-505
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PIPE-505 — Intratympanic injection
  Arms: PIPE-505
Drug: Placebo — Intratympanic injection
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind study of PIPE-505, or placebo, in subjects with hearing loss associated with speech-in-noise impairment.

DETAILED DESCRIPTION:
This is a randomized-controlled, double-blind study of PIPE-505 or placebo given as an injection one time in subjects with sensorineural hearing loss associated with speech-in-noise difficulty. Visits to the clinic will occur at baseline, dosing, and days 1, 7, 14, 30, 60 and 90 after treatment. Safety will be assessed by periodic measurement of vital signs, ear examination, electrocardiogram (ECG), blood laboratory analyses and occurrence of adverse events (AE). Efficacy will be assessed by periodic audiometry and other audiological tests.

ELIGIBILITY:
Inclusion Criteria:

* Subject's primary language is English.
* Male or female between 18 and 75 years of age, inclusive, at randomization.
* Diagnosis of bilateral sensorineural hearing loss (SNHL).
* Normal tympanogram in the ear intended for injection (as defined in protocol) at Screening.
* Male or female subjects with reproductive potential agree to comply with protocol-approved double barrier contraceptive method during and for 3 months after study drug administration.
* The subject is in general good medical health with no clinically significant or relevant abnormalities, including medical history, physical exam, vital signs, ECG, and laboratory evaluations (hematology, chemistry, and urinalysis) as assessed by the Investigator.

Exclusion Criteria:

* History of chronic otitis externa or media, other chronic middle ear disorders, barotrauma, Meniere's disease, endolymphatic hydrops, perilymph fistula, herpes zoster oticus or other infectious etiology of hearing loss.
* Presence of a genetic, syndromal or developmental auditory disorder or of an autoimmune or serious neurological disorder that could contribute to auditory loss.
* Evidence of current conductive hearing loss, mixed hearing loss or otosclerosis.
* History of auditory loss related to exposure to known high-dose ototoxic drugs; any prior exposure to platinum-based medications.
* Otological disorders that would preclude safe tympanic injection.
* Presence of a cochlear implant.
* Evidence of bothersome tinnitus as determined by the Investigator.
* Intratympanic injection within 6 months of randomization.
* Use of an investigational product or intervention other than a non-interventional registry study (including vaccine studies) within the greater of 30 days or 5 half-lives (if known) prior to Screening or expected during the study.
* History of malignancy under current active treatment or considered at substantial risk for progression or recurrence during the study interval, as determined by the Investigator. Note, central nervous system neoplasms or head and neck cancer are excluded from eligibility regardless of treatment status.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Huhn, MD, Study Director — Chief Medical Officer, Pipeline Therapeutics, Inc
Locations (8):
- United States (8):
  - Breathe Clear Institute, Torrance, California
  - ENT and Allergy Associates of Florida, Boca Raton, Florida
  - Advanced ENT & Allergy, New Albany, Indiana
  - University of Kansas; Dept of Otolaryngology Head & Neck Surgery, Kansas City, Kansas
  - Advanced ENT & Allergy, Louisville, Kentucky
  - Charlotte Eye Ear Nose Throat Associates, Charlotte, North Carolina
  - Piedmont Ear Nose Throat and Associates, Winston-Salem, North Carolina
  - Chrysalis Clinical Research, St. George, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Diluent alone: Intratympanic injection
Period: Overall Study
Arm/Group | PIPE-505 | Placebo
Started | 21 | 7
Completed | 21 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PIPE-505 | Placebo | Total
Number analyzed (Participants) | 21 | 7 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (7.93) | 58.9 (11.22) | 62.2 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 3 | 17
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 20 | 7 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 20 | 7 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 7 | 28

OUTCOME MEASURES:

1. Primary Outcome: Safety: Treatment-Emergent Adverse Events (TEAE)
Description: Number of participants with TEAEs
Time Frame: From baseline to 3 months follow up
Measure: Count of Participants; unit: Participants
Arm/Group | PIPE-505 | Placebo
Number analyzed (Participants) | 21 | 7
Participants | 13 | 5

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | PIPE-505 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/7
Other Adverse Events (participants affected / at risk) | 13/21 | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PIPE-505 (N=21) | Placebo (N=7)
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 2 | 0
Ear discomfort (Ear and labyrinth disorders) | 5 | 2
Ear pain (Ear and labyrinth disorders) | 3 | 0
Ear pruritus (Ear and labyrinth disorders) | 2 | 1
Hypoacusis (Ear and labyrinth disorders) | 2 | 1
Inner ear disorder (Ear and labyrinth disorders) | 5 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Tympanic membrane hyperemia (Ear and labyrinth disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 1
Blood glucose increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count increased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 1
Headache (Nervous system disorders) | 1 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT04462198/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT04462198/SAP_001.pdf